CLINICAL TRIAL: NCT00626665
Title: Randomised Control Trial to Assess the Efficacy of Tadalafil in Raynaud's Phenomenon in Scleroderma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanjay Gandhi Postgraduate Institute of Medical Sciences (Other Government)
Responsible Party: Principal Investigator, Vikas Agarwal, Additional Professor, Sanjay Gandhi Postgraduate Institute of Medical Sciences
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: A-15;PGI/DM/EC/40/7/11/07
Record Dates: First submitted 2008-02-21; First posted 2008-02-29 (Estimated); Last update posted 2013-03-22 (Estimated); Status verified 2013-03

CONDITIONS: Raynaud Disease
Keywords: Raynaud disease; Scleroderma
MeSH Terms: conditions — Raynaud Disease; Scleroderma, Diffuse | interventions — Tadalafil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Placebo (Placebo Comparator): One placebo tablet every alternate day for 6 weeks
  Interventions: Drug: Tadalafil

INTERVENTIONS:
Drug: Tadalafil — Tablets Tadalafil, 20 mg, alternate days, 6 weeks
  Other Names: Tadalis

SUMMARY:
In this double-blinded, placebo-controlled, fixed-dose, study patients will be randomly assigned to take placebo or 20 mg tadalafil thrice weekly for 6 weeks. After 6 weeks a wash out period of 2 week will be observed and then the two groups will be switched over to receive the other drug. We planned a priori to include 20 patients. The concomitant medication for treatment of rheumatic disease remained unchanged during the whole study. Patient will undergo clinical and lab evaluation for organ damage for kidney and lungs. ECHO heart will be done at base line to assess the PAH and LV function and repeated at the end of the study. Blood pressure will be recorded at each visit. A physician unaware of the treatment group will record skin score and appearance of new cutaneous ulcers. The primary outcome variables will be frequency and duration of Raynauds attacks, evolution of trophic digital lesions and change in flow mediated dilatation of the brachial artery. Flow mediated dilatation of the brachial artery will be done at baseline 6 and 12 weeks.

DETAILED DESCRIPTION:
Introduction Raynaud's syndrome, which was first described by Maurice Raynaud in 1862, is defined as episodic cold or emotional stress-triggered ischemic vasospasms of the digital arteries and precapillary arterioles. This phenomenon affects 95% of the systemic sclerosis (SScl) patients and may lead to superficial ulcerations and in severe cases can even result in deep tissue necrosis with gangrene. Raynaud's phenomenon (RP) is symptom of a generalised vasculopathy in SScl, which eventually leads to a fibroproliferative arteriopathy. Pulmonary artery hypertension is one of many serious sequelae of this process. Nonpharmacological therapy includes avoidance of cold temperatures, emotional stress, and smoking. Pharmacological therapy with vasodilators such as calcium channel blockers, alpha adrenergic receptor blockers, or angiotensin II receptor antagonists and other agents has been used. Effects of treatments, however, are often inadequate.1 Sildenafil is a selective inhibitor of cGMP specific phosphodiesterase type 5. Besides its established effect in erectile dysfunction, sildenafil provides cGMP-dependent microvascular and macrovascular dilation and, furthermore, were recently shown to exhibit antiproliferative effects.2 There are a few studies in the literature on the efficacy of sildenafil in Raynaud's disease.3-5 It has been shown by these studies and a few case reports that sildenafil may be useful in RP. The limitation of sildenafil is its short t1/2 (4 hours). Tadalafil is more selective and longer acting (17 hours) analogue of sildenafil.6 These PDE 5 inhibitors have been shown to improve endothelial function in diabetic subjects and cold induced vasospasm.7 It is a well known fact that endothelial dysfunction is one of the major pathogenetic mechanisms in scleroderma8. There has been no randomised control trial on the efficacy of tadalafil in RP. There is one study that had shown beneficial effect of Tadalafil in cold induced vasoconstriction in pateints with Raynaud's phenomenon9. So we designed this study to assess the effect of tadalafil on Raynauds phenomenon and endothelial dysfunction in scleroderma. We hypothesise that the tadalafil improves the Raynaud's phenomenon and endothelial dysfunction in scleroderma patients and can act as a disease-modifying agent.

Patients with systemic, scleroderma will be enrolled.

Study Protocol In this double-blinded, placebo-controlled, fixed-dose, study patients will be randomly assigned to take placebo or 20 mg tadalafil thrice weekly for 6 weeks. After 6 weeks a wash out period of 2 week will be observed and then the two groups will be switched over to receive the other drug. We planned a priori to include 30 patients. The concomitant medication for treatment of rheumatic disease remained unchanged during the whole study. Patient will undergo clinical and lab evaluation for organ damage for kidney and lungs. ECHO heart will be done at base line to assess the PAH and LV function and repeated at the end of the study. Blood pressure will be recorded at each visit. A physician unaware of the treatment group will record skin score and appearance of new cutaneous ulcers. The primary outcome variables will be frequency and duration of Raynaud's attacks, evolution of trophic digital lesions and change in flow mediated dilatation of the brachial artery. Flow mediated dilatation of the brachial artery will be done at baseline 6 and 12 weeks.

Clinical Evaluation Symptoms of Raynaud's phenomenon will be assessed by diary cards. When an attack occurred, patients immediately recorded the event and its duration in the diary. At the end of each day, patients gave an overall estimation of the last 24 hours, using a 10-point Raynaud's Condition Score (0 points - subject felt not handicapped by Raynauds attacks; 10 points - subject felt extremely handicapped) validated as described elsewhere. Local Temperature will be recorded in a separate column in the diary daily.

Assessment of cutaneous digital tip ulcers/ infarcts:

The number and position of cutaneous digital tip ulcers or infarcts on any finger will be recorded. Data on both ulcers and infarcts will be collected.

Health Assessment Questionnaire (HAQ):

The HAQ is a self-administered instrument that measures physical disability in 8 domains of function: dressing/grooming, arising, eating, walking, hygiene, reach, grip, and activity. A visual analog scale (VAS) for pain is also part of the HAQ. The results for the 8 subscales, the composite disability score, and the pain measurement are each reported on a 0-3 scale. The HAQ has been used extensively in studies of rheumatoid arthritis and has also been validated in patients with scleroderma. Levels of circulating soluble markers of endothelial cell function, including soluble isoforms of endothelin 1 (ET-1), von Willebrand factor (vWF), and procollagen type I N-terminal propeptide (PINP) will be measured at 0 and 12 weeks Statistics Students T test will be applied to the continuous variables whereas chi square test will be applied to categorical variables.

From an analysis of the daily record sheets, the Following will be calculated: (i) the total average daily duration of the attacks (TADDA), obtained by dividing the total duration in min of attacks during a given three -week interval (observation period) by the number of diary days; (ii) the average duration of a single attack (ADSA), by dividing the overall duration by the number of attacks during the observation period; (iii) the average daily frequency of the attacks (ADFA), by dividing the total number of attacks during the interval considered (3 weeks) by the number of diary days; and (iv) the severity of the attacks, measured on a visual analogical scale; this will be designated the Raynaud's condition score (RCS) and will be calculated as the arithmetic average of the daily scores during the interval considered (3weeks).

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects between the ages of 18 years and 60 years will be selected for the study if they have a clinical diagnosis of Raynaud's phenomenon secondary to systemic sclerosis (scleroderma). Raynaud's phenomenon is defined as a history of cold sensitivity associated with colour changes of cyanosis or pallor, as well as a history of at least 4 attacks per week during two pre-trial period even with treatment with other vasodilators. The diagnosis of scleroderma is defined by the American College of Rheumatology (ACR) criteria or by the presence of at least 3 of the 5 features of the CREST syndrome (calcinosis, Raynaud's phenomenon, esophageal dysmotility, sclerodactyly, telangiectasias).

Exclusion Criteria:

Patients will be excluded if they have:

* Symptomatic orthostatic hypotension
* Evidence of current malignancy
* History of sympathectomy
* Upper extremity deep vein thrombosis or lymphedema within 3 months
* Recent surgical procedure requiring general anesthesia
* AMI, unstable angina, strokes and TIA within the past three months
* Smoking
* Use of any investigational drug within 30 days of the study sessions
* Use of medications that might interfere with tadalafil like nitrates and alpha adrenergic blockers that have vasoactive effects, and patients taking potent inhibitors of CYP3A4 such as ritonavir, ketoconazole, and itraconazole, erythromycin, itraconazole, and grapefruit juice
* Patients taking alcohol
* Patients with bleeding disorders
* Significant active peptic ulceration
* Current pregnancy
* Current breast-feeding

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2007-12; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
The primary outcome variables will be frequency and duration of Raynaud's attacks, evolution of trophic digital lesions | 6 weeeks and 12 weeks

SECONDARY OUTCOMES:
change in flow mediated dilatation of the brachial artery | 6 weeks and 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Vikas Agarwal, MD, DM, Principal Investigator — Sanjay Gandhi Postgraduate Institute of Medical Sciences

REFERENCES:
- [Result] Shenoy PD, Kumar S, Jha LK, Choudhary SK, Singh U, Misra R, Agarwal V. Efficacy of tadalafil in secondary Raynaud's phenomenon resistant to vasodilator therapy: a double-blind randomized cross-over trial. Rheumatology (Oxford). 2010 Dec;49(12):2420-8. doi: 10.1093/rheumatology/keq291. Epub 2010 Sep 12. PMID 20837499